CLINICAL TRIAL: NCT02028091
Title: Diabetes Mellitus - A Diagnosis Trial by Means of Non Invasive Measurements
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Wolfgang SCHRAMM, Ao Univ. Prof. Dr., Medical University of Vienna
Other Study IDs: 1242/2012
Record Dates: First submitted 2014-01-03; First posted 2014-01-06 (Estimated); Last update posted 2014-01-07 (Estimated); Status verified 2014-01

CONDITIONS: Diabetes Mellitus Type II
Keywords: Pulse walve arrival time differences
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Diabetes mellitus: All patients over 18 years with diagnosed diabetes mellitus type II.
- Non Diabetic: Patients over 18 years with no known diabetes mellitus or other known/diagnosed vascular diseases.

SUMMARY:
Vascular damage caused by diabetes mellitus, cigarette smoking, age and arterial hypertension theoretically changes pulse wave velocity.

DETAILED DESCRIPTION:
Diabetes mellitus related vascular alterations are associated with an increased risk of hypertonia, atherosclerosis, neuropathy, diabetic retinopathy, and further more.

Increased vascular rigidity, which is based on the increased stiffness of vessels caused by vascular damage leads to an increase of pulse wave velocity. This assumption is based on the Moens-Korteweg-equation which is calculated using the modus of arterial vessel elasticity, arterial vessel wall thickness, the arterial radius and blood viscosity.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years

Exclusion Criteria:

* Diabetic foot gangrene
* No possibility of pulse wave velocitiy measurement on the finger or toe

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 50 patients over 18 years with diagnosed type II diabetes mellitus are included into the diabetes group.
  50 healthy patients with no known or diagnosed diabetes mellitus or damage of the vessels are included into the non diabetes group.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2012-09; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Pulse wave arrival time difference between finger and toe, duration of diabetes | 1 Minute data recording of the pulse waves at four sites.
  The pulse wave is recorded by plethysmography using a pulse-oximeter and a continuous noninvasive arterial blood pressure measurement (CNAP-500) device, both on the finger and toe. The time between these 4 recorded waves is then calculated. The influence of age, duration of known arterial hypertension, cigarette smoking (pack-years) and diabetes mellitus.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Vienna, Austria

REFERENCES:
- [Background] Alberti KG, Zimmet PZ. Definition, diagnosis and classification of diabetes mellitus and its complications. Part 1: diagnosis and classification of diabetes mellitus provisional report of a WHO consultation. Diabet Med. 1998 Jul;15(7):539-53. doi: 10.1002/(SICI)1096-9136(199807)15:73.0.CO;2-S. PMID 9686693
- [Background] Babchenko A, Davidson E, Adler D, Ginosar Y, Kurz V, Nitzan M. Increase in pulse transit time to the foot after epidural anaesthesia treatment. Med Biol Eng Comput. 2000 Nov;38(6):674-9. doi: 10.1007/BF02344874. PMID 11217886
- [Background] Chen YT, Chiayg CY, Wang MC, Tsai WC, Wu HT, Liu CC. Serial changes of pulse wave velocity and correlations with hemodynamic parameters during general anesthesia. Acta Anaesthesiol Taiwan. 2006 Dec;44(4):193-8. PMID 17233362
- [Background] Chowienczyk PJ, Kelly RP, MacCallum H, Millasseau SC, Andersson TL, Gosling RG, Ritter JM, Anggard EE. Photoplethysmographic assessment of pulse wave reflection: blunted response to endothelium-dependent beta2-adrenergic vasodilation in type II diabetes mellitus. J Am Coll Cardiol. 1999 Dec;34(7):2007-14. doi: 10.1016/s0735-1097(99)00441-6. PMID 10588217
- [Background] Foo JY, Wilson SJ, Williams G, Harris MA, Cooper D. Age-related factors that confound peripheral pulse timing characteristics in Caucasian children. J Hum Hypertens. 2005 Jun;19(6):463-6. doi: 10.1038/sj.jhh.1001846. PMID 15729376
- [Background] Dickersin K, Min YI, Meinert CL. Factors influencing publication of research results. Follow-up of applications submitted to two institutional review boards. JAMA. 1992 Jan 15;267(3):374-8. PMID 1727960
- [Background] Foo JY, Wilson SJ, Williams G, Harris MA, Cooper D. Pulse transit time as a derived noninvasive mean to monitor arterial distensibility changes in children. J Hum Hypertens. 2005 Sep;19(9):723-9. doi: 10.1038/sj.jhh.1001891. PMID 15920454
- [Background] Foo JY, Lim CS. Pulse transit time as an indirect marker for variations in cardiovascular related reactivity. Technol Health Care. 2006;14(2):97-108. PMID 16720953
- [Background] Harris MI. Undiagnosed NIDDM: clinical and public health issues. Diabetes Care. 1993 Apr;16(4):642-52. doi: 10.2337/diacare.16.4.642. No abstract available. PMID 8462395
- [Background] Jaryal AK, Selvaraj N, Santhosh J, Anand S, Deepak KK. Monitoring of cardiovascular reactivity to cold stress using digital volume pulse characteristics in health and diabetes. J Clin Monit Comput. 2009 Apr;23(2):123-30. doi: 10.1007/s10877-009-9174-z. Epub 2009 Mar 24. PMID 19308667
- [Background] Kinsella SM, Whitwam JG, Spencer JA. Aortic compression by the uterus: identification with the Finapres digital arterial pressure instrument. Br J Obstet Gynaecol. 1990 Aug;97(8):700-5. doi: 10.1111/j.1471-0528.1990.tb16242.x. PMID 2400747
- [Background] Kelly RP, Millasseau SC, Ritter JM, Chowienczyk PJ. Vasoactive drugs influence aortic augmentation index independently of pulse-wave velocity in healthy men. Hypertension. 2001 Jun;37(6):1429-33. doi: 10.1161/01.hyp.37.6.1429. PMID 11408390